CLINICAL TRIAL: NCT06765291
Title: Behavioral Intervention for Youth to Promote Vaping Cessation
Acronym: VIA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Anne Eden Evins, Professor of Psychiatry, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 24-560; R01CA287721 (NIH)
Record Dates: First submitted 2025-01-03; First posted 2025-01-09 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Vaping; Vaping Teens; Nicotine Dependence
Keywords: Vaping; Nicotine Depedence; Vaping Cessation
MeSH Terms: conditions — Vaping; Tobacco Use Disorder

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- QuitVaping (QV) (Experimental): Participants will:
  * Attend QuitVaping behavioral support sessions, completed via videoconference or in-person, once per week for 12 weeks
  * Be encouraged to sign up for This is Quitting (TIQ), a text message vaping cessation program for adolescents
  Interventions: Behavioral: QuitVaping; Behavioral: This is Quitting (TIQ)
- Enhanced Usual Care (EUC) (Active Comparator): Participants will:
  * Be encouraged to sign up for This is Quitting (TIQ), a text message vaping cessation program for adolescents
  * Attend no behavioral support sessions
  Interventions: Behavioral: This is Quitting (TIQ)

INTERVENTIONS:
Behavioral: QuitVaping — QuitVaping is a manualized intervention based on the American Lung Association smoking cessation program modified with adolescent appropriate content and language for vaping cessation from the vaping section of teen.smokefree.gov and the Truth Initiative. These behavioral support sessions will be delivered weekly during the 12-week treatment phase via videoconference or in- person.
  Arms: QuitVaping (QV)
Behavioral: This is Quitting (TIQ) — A free, publicly available text message vaping cessation program from Truth Initiative, designed specifically to help adolescents who vape nicotine quit. Participants who set a quit date receive messages for a week preceding it and 30 days afterward that include encouragement and support, skill- and self-efficacy building exercises, coping strategies, and information about the risks of vaping, benefits of quitting and cutting down to quit.

SUMMARY:
This study will test the hypothesis that the QuitVaping (QV) intervention and additional texting support will improve nicotine abstinence rates in adolescents as compared to Enhanced Usual Care (EUC: education about nicotine, vaping and addiction, advice to quit vaping, referral to TIQ texting support). Approximately 400 adolescents will be randomly assigned to one of two arms (1) QuitVaping intervention plus texting support to quit vaping and (2) EUC only.

DETAILED DESCRIPTION:
Up to 400 adolescents, ages 14-18, who report weekly nicotine vaping (or use of other non combusted nicotine products, "vaping") and are willing to try to quit or reduce vaping will be enrolled; eligible participants will be randomly assigned in a 1:1 ratio to a double-blind intervention consisting of (1) QuitVaping intervention plus texting support or (2) EUC only.

Participants assigned to the QuitVaping intervention will receive referral to TIQ texting app and 12 brief, weekly, study intervention visits with monthly follow up visits until week 36. Those who are assigned to EUC will be offered TIQ texting app referral to support vaping cessation. All participants will receive education about nicotine, vaping and addiction, advice to quit vaping, TIQ referral, and weekly blinded assessments with biochemical verification of abstinence. The person conducting the assessment will be blind to study condition such that the intervention will be double blind. Following completion of the 12-week intervention period, participants will have follow-up visits at weeks 16, 20, 24, 28, 32, and 36. Visits will be conducted remotely on a secure video conferencing platform or in-person.

The enrollment visit will include a detailed description of the study, informed consent/assent, assessments to confirm eligibility, assessments of vaping and other drug use behavior, and medical and psychiatric diagnostic and symptom assessments. Written informed consent will be obtained from participants age 18 years. An opt-out consent form will be sent to a parent or legal guardian of participants ages 14-17. If a parent or legal guardian does not opt their child out within two weeks of verified review of the opt out consent form, the participant is considered consented and written informed assent will be obtained.

Eligible, consented participants will then be scheduled for weekly visits which will include assessments for all participants, and behavioral vaping cessation sessions for those assigned to QuitVaping. Saliva will be collected at assessment visits for cotinine measurement in participants who report nicotine abstinence. Urine NNAL will be collected at week 12 in participants who report continuous 4-week abstinence (weeks 9-12). Instructions for how to perform the tests will be sent to participants, and during virtual assessment visits, participants will hold the assays up to their device's camera so study staff can record the test results.

ELIGIBILITY:
Inclusion Criteria:

* Age 14-18 inclusive
* Self-report of at least weekly nicotine vaping (or use of other non combusted nicotine products, "vaping") for the prior ≥3 months
* Self-report of no regular combusted tobacco use (i.e., 5 or more days of smoke smoked tobacco use per week) prior to enrollment and exhaled CO <10 ppm for those with an in person baseline visit
* Report willingness to try to quit or reduce vaping in the next 30 days
* Able to understand study procedures and read and write in English or Spanish
* Have a parent or legal guardian who is able to participate in the opt out process
* Competent and willing to provide written informed consent (if age 18) or assent (if under 18)

Exclusion Criteria:

* Use of a smoking cessation medication in the prior month (nicotine patch, gum, nasal spray, or inhaler, varenicline, bupropion)
* Unwilling to abstain during the study from using smoking cessation aids other than those provided by the study
* Unwilling to provide saliva or urine samples
* Any condition or situation that would, in the investigator's opinion, make it unlikely that the participant could adhere safely to the study protocol

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-06-18 (Actual); Primary Completion 2028-03-29 (Estimated); Study Completion 2028-09-27 (Estimated)

PRIMARY OUTCOMES:
Continuous 4-week nicotine vaping abstinence at end of treatment | From week 9 to week 12
  The percent of participants who self-report nicotine vaping abstinence since the last visit on the timeline followback interview and have cotinine <10ng/mL, assessed at study weeks 9-12. The primary comparison of interest is between the QV + EUC arms.

SECONDARY OUTCOMES:
Continuous continine-verified nicotine vaping abstinence at the end of follow up (Weeks 9-36) | From week 9 to week 36
  The percent of participants who self-report nicotine vaping abstinence since the last visit on the timeline followback interview and have cotinine <10ng/mL, assessed at study weeks 9-36. The primary comparison of interest is between the QV + EUC arms.

CONTACTS AND LOCATIONS:
Overall Officials: A. Eden Evins, MD, MPH, Principal Investigator — Massachusetts General Hospital; Randi M. Schuster, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Center for Addiction Medicine, 101 Merrimac Street, Suite 320, Boston, MA 02114, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD will be deposited in the NIMH Data Archive. This is a free data repository open to qualified researchers from all mental health and other research communities to share, archive, cite, access, and explore research data. Clinical data necessary to validate and replicate research findings, including questionnaires, interviews, and saliva cotinine test results will be shared.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Scientific data will be available one year after the grant end date specified on the first Notice of Award. Scientific data included in published manuscripts will be made available at the time of publication. Scientific data and the code/software/tools used to development the published or submitted dataset will be shared at the time of data submission or publication and maintained for no shorter than five years.
Access Criteria: Data access will be controlled. In order to access shared data, qualified researchers will be required to complete a data use certification and receive approval from NDA Data Access Committee.